CLINICAL TRIAL: NCT00871637
Title: Airway Macrophages and Sputum Milieu in Adult Subjects With Airflow Obstruction
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0222-08-FB
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Occupational Diseases; Tobacco Use Disorder
Keywords: Pulmonary disease, chronic obstructive; Airway macrophages; Sputum milieu; Airway inflammation; Occupational diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Occupational Diseases; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group One: Healthy non-smoking controls
- Group Two: Smoking adults with chronic bronchitis/chronic obstructive pulmonary disease
- Group Three: Non-smoking adults with chronic bronchitis/chronic obstructive pulmonary disease

SUMMARY:
Airway macrophage impairment is a central feature in the immunopathogenesis of chronic obstructive pulmonary disease, regardless of smoking status.

DETAILED DESCRIPTION:
In the United States, a variety of farming operations can generate significant amounts of dust. Chronic organic dust exposure to workers in this industry can result in several respiratory health conditions including chronic bronchitis, chronic obstructive pulmonary disease (COPD), and exacerbations of asthma. Organic dust is a complex mixture containing particulate matter and microbial-associated components from gram positive and gram negative bacteria. Airway macrophages are key innate immune cells that are rapidly activated by exposure to inhaled toxins and organic dust.

The literature indicates that subjects with tobacco-induced chronic bronchitis/COPD have alveolar macrophages that have impaired function. It has been hypothesized that the impaired lung macrophage function may contribute to the increased susceptibility to infections and chronic bacterial colonization that is a central feature in subjects with chronic bronchitis/COPD. It is unknown at this time if impaired macrophage function is secondary to tobacco-induced effects, or is a central pathologic feature of chronic bronchitis/COPD.

We will explore the expression of innate immune cell surface molecule expression involved in antigen presentation, phagocytic ability, and ex vivo cytokine responses in airway macrophages obtained by induced sputum. We will also collect blood to determine if ex vivo stimulation of blood mimics the inflammatory responses observed with airway macrophages. Comparisons to our past findings in vitro studies, which demonstrated that repetitive organic dust exposure impairs monocyte derived macrophage immune cell surface markers and function, could then be made. This information could lead to future investigations centered on therapeutic interventions to prevent or reverse the underlying lung disease experienced by farmers in this industry.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable to participate in induced sputums
* Group One: Smoked less than 100 cigarettes in their lifetime Quit smoking greater than 10 years ago Pre-bronchodilator FEV1/FVC > 70% Pre-bronchodilator FEV1 % predicted > 80%
* Group Two: Greater than a 20-pack year tobacco history Smoked in the last two years Post-bronchodilator FEV1/FVC < 70%
* Group Three:Have less than a 20-pack year tobacco history Quit smoking greater than 20 years ago Post-bronchodilator FEV1/FVC < 70%

Exclusion Criteria:

* Personal history of lung cancer
* Pregnancy
* Personal history of autoimmune disease
* Currently taking oral/parental corticosteroids
* Personal history of upper or lower respiratory tract infection in the prior four weeks

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups Group One : Healthy non-smoking controls Group Two : Smoking adults with chronic bronchitis/COPD Group Three: Non-smoking adults with chronic bronchitis/COPD
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of airway macrophages for immune cell surface marker expression and phagocytic ability in adults with airflow obstruction & healthy controls | One year
  Determine if airway macrophages from adult participants with airflow obstruction demonstrate impaired innate immune cell surface marker expression and phagocytic ability compared to healthy controls.

SECONDARY OUTCOMES:
Comparison of airway macrophages for cytokine responsiveness in adults with airflow obstruction & healthy controls | One year
  Determine if airway macrophages from adult participants with airflow obstruction demonstrate impaired cytokine responsiveness compared to healthy controls.
Comparison of airway macrophage cytokine responsiveness to whole blood cytokine responsiveness | One year
  Determine if airway macrophage cytokine responsiveness is comparable to whole blood cytokine responsiveness.
Determining if immunomodulators in airway sputum milieu f predict airway macrophage phenotype and function | One year
  To determine if airway sputum milieu for potential immunomodulators predict airway macrophage phenotype and function.

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Poole, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska, Omaha, Nebraska, United States

REFERENCES:
- [Result] Harting JR, Gleason A, Romberger DJ, Von Essen SG, Qiu F, Alexis N, Poole JA. Chronic obstructive pulmonary disease patients have greater systemic responsiveness to ex vivo stimulation with swine dust extract and its components versus healthy volunteers. J Toxicol Environ Health A. 2012;75(24):1456-70. doi: 10.1080/15287394.2012.722186. PMID 23116451